CLINICAL TRIAL: NCT06314997
Title: Dynamic Changes in RAS Gene Status and HER2 Expression in Circulating Tumour Cells: a Phase II Trial
Brief Title: Dynamic Changes in Circulating Tumour Cells Protein Expression
Acronym: Liquid-DRER2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Matteo's Friends (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2013.34
Record Dates: First submitted 2024-02-13; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Recurrence Free Survival
MeSH Terms: interventions — Panitumumab

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RAS unmutated CTCs HER positive (Experimental)
  Interventions: Drug: panitumumab (EGFR inhibitors)
- CTCs (Experimental)
  Interventions: Drug: panitumumab (EGFR inhibitors)
- RAS unmutated CTCs HER negative (Experimental)
  Interventions: Drug: panitumumab (EGFR inhibitors)

INTERVENTIONS:
Drug: panitumumab (EGFR inhibitors) — Chemotherapy treatment includes anti-EGFR biologics such as cetuximab or panitumumab, antiangiogenic drugs such as bevacizumab or aflibercept. The indication to treat depends from the presence of CTCs analysed for Ras mutation and HER2 expression

SUMMARY:
This multicenter study, randomized, controlled of blood-based biomarker-driven targhet therapy. Patients were selectedm( at Hospital San Giovanni and Celio in Rome) according to CTCs results ( CTCs-guided managment performed at University Magna Graecia) or managed by the treating clinician according to standard pathological criteria (standard management). The participants were assigned to trial groups with the use of block randomization stratified according to the enrolling center location metropolitan) and tumor stage (T3 or T4).

DETAILED DESCRIPTION:
The investigators enroll patients with histologically confirmed advanced stage (T3 or T4, N1/2, M0/1) colorectal adenocarcinoma with molecular analysis on RAS mutant status. The participants are enrolled within 3 weeks at the time of progression disease (PD) from any line of therapy. Blood samples were collected from each participant after obtaining informed consent. Permission to perform CTCs analysis from blood was obtained from the Regional Ethical Committee (No.2013/34) and the study is conducted in accordance with the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance-status score of 0 to 2 (scores range from 0 to 5, with higher numbers reflecting greater disability) ,
* medically able to receive chemotherapy.

Exclusion Criteria:

* evidence of infective disease before enrollment ,
* a history of another primary cancer within the previous 3 years,
* the presence of synchronous primary colorectal cancer.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-01-14 (Actual); Primary Completion 2024-12-17 (Estimated); Study Completion 2027-12-18 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy end point was recurrence- free survival at 12 months. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Natalia Malara, Germaneto, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malara N, Donato G, Ferrazzo F, Garo NC, Fulciniti F. The Charactex Protocol for Blood-Derived Cytological Preparation of Nonhematological Cancer. Acta Cytol. 2023;67(3):295-303. doi: 10.1159/000527904. Epub 2022 Dec 12. PMID 36509041
- [Background] Malara N, Coluccio ML, Grillo F, Ferrazzo T, Garo NC, Donato G, Lavecchia A, Fulciniti F, Sapino A, Cascardi E, Pellegrini A, Foxi P, Furlanello C, Negri G, Fadda G, Capitanio A, Pullano S, Garo VM, Ferrazzo F, Lowe A, Torsello A, Candeloro P, Gentile F. Multicancer screening test based on the detection of circulating non haematological proliferating atypical cells. Mol Cancer. 2024 Feb 13;23(1):32. doi: 10.1186/s12943-024-01951-x. PMID 38350884
- [Background] Malara N, Trunzo V, Foresta U, Amodio N, De Vitis S, Roveda L, Fava M, Coluccio M, Macri R, Di Vito A, Costa N, Mignogna C, Britti D, Palma E, Mollace V. Ex-vivo characterization of circulating colon cancer cells distinguished in stem and differentiated subset provides useful biomarker for personalized metastatic risk assessment. J Transl Med. 2016 May 12;14(1):133. doi: 10.1186/s12967-016-0876-y. PMID 27176720